CLINICAL TRIAL: NCT04277715
Title: Development of a Parent Training Intervention for Pediatric Patients With Medically Unexplained Symptoms
Brief Title: Parent Training for Youth With Chronic Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: The Wallace Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2000027265
Record Dates: First submitted 2020-02-17; First posted 2020-02-20 (Actual); Last update posted 2023-09-14 (Actual); Status verified 2023-09

CONDITIONS: Medically Unexplained Symptoms
MeSH Terms: conditions — Medically Unexplained Symptoms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Parent training (Experimental): Parents of participating children with chronic symptoms will receive the intervention in a virtual group format. Groups will last 90-minutes and run for 6-8 weeks. Groups will be co-led by a clinical psychologist and pediatric physician with expertise in child behavioral interventions and medically unexplained symptoms.
  Interventions: Behavioral: Parent training

INTERVENTIONS:
Behavioral: Parent training — Parents will learn evidence-based techniques for increasing support and decreasing accommodation of children's chronic symptoms.

SUMMARY:
The purpose of this study is to examine the effects of a parent-only, group-based intervention intended to treat youth with chronic, unexplained medical symptoms such as (but not limited to) chronic fatigue, musculoskeletal pain, headache, and abdominal pain. Prior to and following the intervention, the child and parent(s) will be asked to complete several questionnaires about their well-being and functioning. The investigators predict that participation in this intervention will lead to change in relevant outcomes, including youth symptoms and functional impairment, and parenting stress and accommodation of symptoms. The investigators also predict that this group will be acceptable and feasible for parents.

ELIGIBILITY:
Inclusion Criteria:

* Presence of medically unexplained symptoms, including: fibromyalgia, chronic fatigue, chronic Lyme disease, irritable bowel syndrome, musculoskeletal pain, headache, abdominal pain and related bowel dysfunction, perceived cognitive impairment, or other nonspecific symptoms
* Symptoms must have been present for at least 3 months, associated with some degree of impairment (e.g., missing school), and not attributable to a known organic or medical disorder despite adequate evaluation
* Participants must be proficient or fluent in English
* Children must live with their participating parent(s) at least 50% of the time

Exclusion Criteria:

* Presence of a serious medical condition by history, including chronic autoimmune or inflammatory condition
* Lifetime history of a psychotic disorder, bipolar disorder, Autism, or intellectual disability (Note: this criterion applies to child and parent(s))
* Presence of severe emotional or behavioral problems that require a more immediate treatment

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 16 (Actual)
Dates: Start 2021-04-05 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
Client Satisfaction Questionnaire (CSQ-8; Attkisson & Greenfield, 1996) | Post-treatment (6-8 weeks)
  The CSQ-8 is an 8-item self-report questionnaire that assesses satisfaction with (i.e., acceptability of) services received. Questions are rated on a response scale of 1("Quite dissatisfied") to 4("very satisfied"). An overall score is calculated by summing the respondent's score for each scale item. Scores range from 8 to 32, with higher values indicating higher satisfaction with/acceptability of treatment.

SECONDARY OUTCOMES:
Functional Disability Inventory (FDI; Kashikar-Zuck et al., 2011) | Pre-treatment; Post-treatment; 3-month follow-up
  The FDI is a 15-item rating scale that assesses functional disability (i.e., physical and psycho-social functional impairment) in children and adolescents with chronic pain and related conditions. The FDI has a parent form and a child/adolescent form. Items are rated on a scale of 0 ("No trouble") to 4 ("Impossible"). Total scores range from 0-60, with higher scores indicating greater functional disability, categorized as No/Minimal (0-12), Moderate (13-29), and Severe (30) Disability.
Pediatric Quality of Life Inventory (PedsQL; Varni, Seid, & Kurtin, 2001) | Pre-treatment; Post-treatment; 3-month follow-up
  The PedsQL is a modular, youth- and parent-report questionnaire assessing health-related quality of life in children and adolescents ages 2 to 18. The PedsQL Generic Core Scales contain 23-items about quality of life in physical, emotional, social, and school domains. Response options are on a five-point scale, ranging from 0 ("never") to 4 ("almost always"). Items are summed and higher scores indicate higher well-being.
The Symptom Impact Questionnaire-Revised (SIQR; Bennett, Friend, Jones, Ward, Han, & Ross, 2009) | Pre-treatment; Post-treatment; 3-month follow-up
  The SIQR is used to measure physical function, overall impact of the syndrome, and symptom severity in youth (self- and parent-report). Respondents are asked to rate items on scales such as "no difficulty" to "very difficult" (physical function), "never" to "always" (impact of the syndrome), or "no pain" to "unbearable pain" (example of symptom severity). Total scores range from 0 (indicating no symptom impact) to 100 (extreme symptom impact). A 14% change in scores has been empirically determined to represent minimal clinically significant difference following treatment.
Clinical Global Impression Scale (CGI; National Institutes of Mental Health, 1985) | Pre-treatment; Post-treatment
  The CGI is a clinician-rated measure that assesses overall severity (CGI-S) and improvement (CGI-I) of child symptoms following treatment. CGI-S scores range from 1 ("normal, not at all ill") to 7 ("extremely ill"). CGI-I scores of 1 ("very much improved") or 2 ("much improved") indicate a positive treatment response; all other responses (3 "minimally improved" to 7 "very much worse") are considered negative responses to treatment.
Screen for Child Anxiety Related Emotional Disorders (SCARED; Birmaher, Khetarpal, Brent, Cully, Balach, Kaufman, & Neer, 1997) | Pre-treatment; Post-treatment; 3-month follow-up
  The SCARED is a 41-item self- and parent-report questionnaire assessing a range of anxiety symptoms. It is appropriate for children and adolescents ages 8-18. Items are rated on a 3-point scale ranging from 0 ("not true or hardly ever true") to 2 ("very true or often true"). Items are summed and total scores above 25 indicate the likely presence of an anxiety disorder.
Children's Depression Inventory (CDI-2; Kovacs, 2011). | Pre-treatment; Post-treatment; 3-month follow-up
  The CDI-2 is a 28-item questionnaire assessing depressive symptoms. There are child- and parent- report versions. Respondents are asked to rate symptoms they have experienced (or observed, for parents) over the past two weeks. Each item contains 3 statements scored in order of increasing severity from 0 to 2. Higher total scores indicate greater depressive symptoms.
Family Accommodation Scale - Anxiety (FASA; Lebowitz et al., 2013; Lebowitz, Marin, & Silverman, 2019) | Pre-treatment; Post-treatment; 3-month follow-up
  The FASA is a 13-item parent- and child-report scale that assesses family accommodation of a child's anxiety symptoms. The FASA asks respondents to rate the frequency of parental accommodation, the participation of parents in child's symptoms, and the changes that parents make in routines and schedules due to child's somatic symptoms. Items are rated on a 5-point response scale. Together, these items generate the total accommodation score, with higher scores indicating greater frequency and intensity of accommodation. One additional item assesses the degree of distress the accommodation causes the parents/child, and 4 additional items assess the short-term, negative consequences of not accommodating.
Parenting Stress Index, 4th Edition, Short-Form (PSI-4-SF; Abidin, 2012) | Pre-treatment; Post-treatment; 3-month follow-up
  The PSI-4-SF is a 36-item parent-report scale that assesses three domains of parenting stress, including Parental Distress, Parent-Child Dysfunctional Interaction, and Difficult Child, which combine to form a Total Stress scale. Items are rated on a 5-point scale ranging from 1 ("strongly disagree") to 5 ("strongly agree"), with higher scores indicating more parenting stress.
The Client Credibility Questionnaire (CCQ; Borkovec & Nau, 1972) | Following 1st group session (1 week)
  The CCQ will be used to assess parent expectancies about treatment. To do so, it will be administered to all parents at the end of the first intervention session, after the treatment rationale has been presented. Parents will be asked to make ratings using a scale of 0 to 2 (None, Some, A lot) about: (1) how logical the treatment seems; (2) how confident they are the treatment will be successful, and (3) how confident they would be in recommending the treatment to a friend.
Inventory of Parent Accommodations of Children's Symptoms (IPACS; Harrison, Peterson, Short, & Wetterneck, 2016) | Pre-treatment; Post-treatment; 3-month follow-up
  The ICPACS is a 12-item parent-report measure that assesses the frequency of family accommodation of the child's pain in the past week. Items are rated on a scale ranging from 1 to 5. It includes three subscales: Modifications, Assistance, and Supportive Behaviors. An initial validation study indicated high internal consistency for the total scale (Harrison et al., 2016).
Child's Report of Parental Behavior Inventory (CRPBI; Schludermann & Schludermann, 1988) | Pre-treatment; Post-treatment; 3-month follow-up
  The CRPBI is a 30-item scale used to assess current level of perceived parental behaviors, including acceptance and psychological control. Items are rated on a scale from 1 (Not like…) to 3 (A lot like … my mother). A higher score indicates higher perceived behaviors. There is also a parent-report version of this scale (PRPBI).
Perceived Stress Scale (PSS: Cohen, Kamarck, Mermelstein, 1983) | Pre-treatment; Post-treatment; 3-month follow-up
  The PSS is a 14-item scale that assesses perceived stress of life situations in adolescents and adults. Items are scored on a 5-point scale (0=never to 4=very often). Higher total scores indicate greater levels of perceived stress. The PSS has satisfactory reliability and has well-established validity in relation to physiological stress responses and anxiety and depressive disorders.
Child Anxiety Sensitivity Index (CASI; Silverman, Fleisig, Rabian, & Peterson, 1991) | Pre-treatment; Post-treatment; 3-month follow-up
  The CASI is an 18-item child self-report measure that assesses the extent to which children interpret anxiety symptoms as having negative physical, mental and social consequences. The scale has good construct validity, internal consistency and test-retest reliability (Silverman et al., 1991).
Affective Reactivity Index-Child and Parent versions (ARI-C/P; Stringaris, Goodman, Ferdinando, Razdan, Muhrer, Leibenluft, & Brotman, 2012) | Pre-treatment; Post-treatment; 3-month follow-up
  The ARI-C/P is a parent- and child report measure that assesses frequency, duration, and threshold of child irritability symptoms over 6 months. The ARI-C/P contains 6 items that are rated along a 3-point scale (0 = not true, 1 = somewhat true, 2 = certainly true); total scores range from 0-12. A 7th item, not calculated in the total score, assesses level of general impairment caused by the irritability. The ARI-C/P has shown satisfactory internal consistency, discriminant validity, and is adequately described by a one-factor solution in confirmatory factor analyses.

CONTACTS AND LOCATIONS:
Overall Officials: Wendy Silverman, Ph.D., Principal Investigator — Yale University
Locations (1):
- Yale Child Study Center, Yale University School of Medicine, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No